CLINICAL TRIAL: NCT05128539
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of Recombinant Humanized Anti-PCSK9 Monoclonal Antibody (JS002) Combined With Toripalimab in Patients With Advanced Cancer
Brief Title: A Study Explore JS001+JS002 in Patients With Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The regimen of JS002 75~300mg Q3W has been completed, and the combination therapy is well tolerated and safe. However, considering that the efficacy did not reach the preset, it is recommended to terminate the trial in advance.
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS001-046-I
Record Dates: First submitted 2021-10-27; First posted 2021-11-22 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2021-10

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JS001(Toripalimab)+JS002 (Experimental)
  Interventions: Drug: JS001(Toripalimab)+JS002

INTERVENTIONS:
Drug: JS001(Toripalimab)+JS002 — Part A: In this phase, 3 dose levels will be preliminarily set up. The dose level of Toripalimab is fixed as 240 mg, intravenous infusion, Q3W. The dose levels of JS002 are fixed at 75 mg,150 mg and 300 mg subcutaneously, and the traditional 3+3 design will be used for dose escalation with 21 days as entire treatment cycle. In addition, the period of 21 days after the first administration is defined as the DLT observation period.
  Part B: Based on the data of the safety, PK and preliminary efficacy in Part A patients, the dosage will be determined for advanced tumor patients who had received at least first-line therapy in this part. Two to three groups with different tumor types will be further enrolled, and about 30 patients will be included in each group (the specific number and cohort will be adjusted according to the research progress). Toripalimab is a humanized IgG4κ mAb specific against human PD-1.

SUMMARY:
This open-label phase I clinical study with clinical development phase will evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of JS002 combined with Toripalimab in advanced cancer patients, who has failed standard therapy OR could not tolerate standard therapy OR refused/had no standard therapy.

This study is divided into two parts:

Part A. JS002 combined with Toripalimab dose escalation and dose expansion phase; Part B.JS002 combined with Toripalimab clinical expansion phase.

ELIGIBILITY:
Inclusion criteria:

1. Fully understand and be willing to provide written informed consent;
2. Male or female with age ≥ 18 years and ≤75 years (At part B age ≥18 years);
3. The expected survival is ≥ 3 months;
4. ECOG PS 0 or 1;
5. Advanced tumor patients who have failed standard treatment (including PD-1/PD-L1), cannot tolerate standard treatment, OR refused/have no standard treatment (note: Patients with hepatocellular carcinoma, lung cancer and urothelial carcinoma that have failed PD-1 or PD-L1 treatment are preferred, and other types of the advanced tumor patients without standard treatment can be enrolled according to initial efficacy);
6. Having at least one measurable disease per RECIST 1.1.
7. Agree to provide tumor tissue samples (fresh biopsy samples before treatment should be provided as far as possible; for patients who cannot provide fresh biopsy samples before treatment, archived samples can be provided within 2 years; for some patients who cannot provide qualified tumor tissue samples, they can also be included in the group after discussion and agreement between the investigator and the sponsor);
8. The results of laboratory tests during the screening period indicate that the patient has good organ function:

   a) Hematology (no blood transfusion within 14 days and no treatment with blood components or granulocyte colony cytokines): i. Absolute neutrophil count ANC ≥ 1.5×109/L(1,500/mm3) ii. Platelets ≥ 100×109/L(Part B: ≥ 75×109/L) (100,000/mm3) iii. Hemoglobin ≥ 10.0g/dL (Part B: ≥ 9.0g/dL) b) Hepatic function: i. Serum total bilirubin(TBil) ≤1.5×ULN ; For patients with primary liver cancer, liver metastasis, or proven/suspected Gilbert's disease, TBil ≤ 2×ULN ii. AST and ALT ≤2.5 × ULN; ≤5×ULN in those with hepatic metastasis or primary liver cancer.

   c) Renal function: i. Creatinine clearance(CrCl) ≥50mL/min(Cockcroft-Gault formula); ii. Urine protein ≤ 2+ (if the urine protein is 2+, the 24-h urine protein test will be performed, and only patients with ≤2g are eligible).

   d) Coagulation function: International standardized ratio (PT/INR) and activated partial thrombin time (APTT) ≤1.5×ULN (for those receiving anticoagulant therapy, such as low molecular weight heparin or warfarin, the anticoagulant dose is required to be stable for at least 4 weeks without dose adjustment, and the coagulation parameters INR and APTT at screening are within the expected range of anticoagulant therapy) e) Endocrine function: Thyroid stimulating hormone (TSH) normal, or abnormal TSH but normal FT3 and/or FT4 (for patients with hypothyroidism with abnormal TSH but normal FT4) f) Cardiac function: QTc interval ≤ 460 ms for male and ≤ 480 ms for female, which is calculated according to Fridericia formula.
9. Men or women patients of childbearing potentials agree to use an effective method of contraception (e.g., oral contraceptives, intrauterine devices, or barrier contraception combined with spermicide) and continued to use contraception for 6 months after treatment.
10. Good compliance and follow-up.

Exclusion criteria:

1. A history of malignancies other than the tumors described in this study within 5 years, with the exception of early malignancies that have been completely cured (no recurrence within 5 years), including but not limited to adequately treated thyroid cancer, carcinoma in situ of the cervix, basal or squamous cell skin cancer, and ductal carcinoma in situ after the radical mastectomy);
2. The patients received systemic antitumor drugs(chemotherapy, small molecular targeted drug therapy, hormone therapy, immunotherapy or biological treatment, etc.), local anti-tumor therapy (e.g., patients accepted palliative radiotherapy for bone metastases are eligible, in which the radiotherapy is performed more than 2 weeks before the baseline tumor assessment ), or clinical research drug/treatment instrument within 4 weeks prior to first dose;
3. Patients who have previously received PCKS9 inhibitor therapy;
4. Adverse reactions caused by previous treatment have not recovered to GRADE 1 or below per CTCAE (version 5.0) (except alopecia and neurotoxicity, which investigator judged could not be recovered for a long time);
5. Previous allogeneic hematopoietic stem cell transplantation or solid organ transplantation;
6. Having untreated central nervous system metastasis, or meningeal metastasis. Patients who has received treatment for brain metastases are eligible if meet all the following criterion; stable condition is observed at least 3 months; no radiological progression is identified within 4 weeks prior to first dose; all the nervous system symptoms have returned to baseline levels; no new evidence or expanded brain metastases; has stopped radiotherapy, surgery or steroid therapy at least 28 days prior to first dose;
7. Autoimmune diseases, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, etc., diagnosed within 2 years are ineligible, except for type I diabetes controlled by replacement therapy, skin diseases that do not require systemic treatment (e.g., psoriasis and vitiligo), endocrine diseases controlled by hormone replacement therapy (e.g., hypothyroidism);
8. Patients with associated clinical symptoms (dyspnea, wheezing, abdominal distension, etc.), uncontrolled or repetitive drainage of pleural/abdominal effusion or pericardial effusion. The patients with pleural/abdominal effusion are not allowed to accept intrapleural/intraperitoneal injection of anti-tumor agents accordingly;
9. Have serious cardiovascular and cerebrovascular diseases, such as poorly controlled hypertension (systolic blood pressure > 150mmHg and/or diastolic blood pressure > 100mmHg) or pulmonary hypertension as judged by the investigator; Unstable angina or myocardial infarction, coronary artery bypass grafting or stenting within 6 months prior to study use; Chronic heart failure with heart function grade 2 or greater (NYHA); Degree ⅱ or higher heart block; Grade ≥2 supraventricular or ventricular arrhythmias; Left ventricular ejection fraction (LVEF) < 50%; Cerebrovascular accident (CVA) or transient ischemic attack (TIA) occurred within 6 months prior to medication;
10. History of pulmonary disease: drug-induced interstitial lung disease or pneumonia, obstructive pulmonary disease that severely affects lung function, and symptomatic bronchospasm;
11. Has an active infection requiring systemic treatment;
12. Human immunodeficiency virus (HIV) antibody test positive;
13. Patients with non-alcoholic steatohepatitis, alcoholic/drug-related/autoimmune hepatitis or uncontrolled active hepatitis B virus (HBV), or hepatitis C virus (HCV):

    1. Active HBV infection is defined as patients with surface antigen (HBsAg) positive and detectable DNA higher than the upper limit of the reference in each research center, accompanied with increased ALT; active HCV infection is defined as patients with positive HCV antibody and positive HCV RNA.
    2. Patients with active HBV can take antiviral drugs, such as nucleoside (acid) analogues (NAs), as recommended in the Guidelines for the Prevention and Treatment of Chronic Hepatitis B (2019 edition). Prior to the first dose, patients with HBV DNA < 2000 IU/ mL can participate in this study.
    3. Patients who test positive for HCV antibodies can only be enrolled in this study if the polymerase chain reaction (PCR) test is negative for HCV RNA. D) If the patients were receiving antiviral therapy at the time of enrollment and were required to maintain stable antiviral therapy throughout the study, any patients with compliance concerns were excluded from enrollment.
14. Active tuberculosis (TB) is known to exist. Patients suspected of having active TB should be examined for chest X-rays, sputum cytology, and clinical signs and symptoms.
15. Received systemic corticosteroids (prednisone > 10mg/ day or equivalent) or other immunosuppressive drugs within 14 days prior to the first dose;
16. Have received broad-spectrum antibiotics that may affect gut microbiota within 14 days prior to the first administration;
17. Receiving live or attenuated live vaccine within 4 weeks prior to the first administration;
18. Major surgical procedures (as defined by the investigator, e.g., open biopsy and severe trauma) were performed within 4 weeks prior to the first dose. Note: Intravenous drip replacement is acceptable. Patients who plan to accept major surgery within 30 days after the first dose or not yet fully recovered from previous surgery. Patients with local surgery (e.g., core needle biopsy and prostate biopsy) performed at least 24 h before the first administration are eligible;
19. Those who have a history of psychotropic drug abuse and cannot get rid of it or have a history of mental disorders;
20. Pregnant or lactating women;
21. Patients are allergic to JS002 or Toripalimab and their active ingredients or excipient;
22. Other severe, acute or chronic medical or psychiatric conditions or laboratory abnormalities that, in the investigator's judgment, may increase the risk associated with study participation or may interfere with the interpretation of study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
adverse events (AE)、SAE、irAE | 3 years
  Safety endpoints: adverse events (AE), serious adverse events (SAE), and immune-related adverse events (irAE);
Dose-limiting toxicities (DLTs) | 3 years
  Safety endpoints
MTD | 1 year
  Maximum tolerated dose (MTD)
Recommended dose for extension (RDE) | 1 year
  Recommended dose for extension (RDE)

SECONDARY OUTCOMES:
ORR | 2 years
  Efficacy endpoints: Objective response rate (ORR) based on RECIST 1.1 criteria
DOR | 2 years
  Efficacy endpoints: Uration of response (DOR) based on RECIST 1.1 criteria
DCR | 2 years
  Efficacy endpoints: Disease control rate (DCR) based on RECIST 1.1 criteria
TTR | 2 years
  Efficacy endpoints:Time to response (TTR) based on RECIST 1.1 criteria
PFS | 2 years
  Efficacy endpoints:progression-free survival (PFS) based on RECIST 1.1 criteria
OS | 2 years
  Efficacy endpoints:overall survival (OS) based on RECIST 1.1 criteria
1-year OS rate | 1 year
  Efficacy endpoints: 1-year OS rate based on RECIST 1.1 criteria
Pharmacokinetic (PK) characteristics | 2 years
  Drug concentration of individual subjects at different time points after administration;
Peak concentration（Cmax） | 2 years
  The pharmacokinetic parameters of JS002 and Toripalimab (JS001) :peak concentration (Cmax) ;
Peak time（Tmax） | 2 year
  The pharmacokinetic parameters of JS002 and Toripalimab (JS001) ：peak time (Tmax) ;
Area under blood concentration-time curve (AUC0-T and AUC0-) | 2 years
  The pharmacokinetic parameters of JS002 and Toripalimab (JS001) :area under blood concentration-time curve (AUC0-T and AUC0-) ;
Clearance rate (CL) | 2 years
  The pharmacokinetic parameters of JS002 and Toripalimab (JS001) ：clearance rate (CL) ;
Volume of distribution (Vss) | 2 years
  The pharmacokinetic parameters of JS002 and Toripalimab (JS001) ：volume of distribution (Vss)
Elimination half-life (T1/2) | 2 years
  The pharmacokinetic parameters of JS002 and Toripalimab (JS001) ：elimination half-life (T1/2)
ADA against | 2 years
  Incidences of ADA against JS002 and Toripalimab (JS001), respectively

OTHER OUTCOMES:
Correlation between biomarkers and clinical efficacy | 2 years
  correlation between pD-L1 expression in tumor tissues and efficacy; Analysis of tumor mutation load (TMB) and Tumor microsatellite instability (MSI) in tumor tissues and paired blood samples by whole exon sequencing (WES),Peripheral blood immune cell surface receptor (PD-1, MHC-I expression level) detection

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Tumor Hospital, Zhengzhou, Henan, China